CLINICAL TRIAL: NCT02176720
Title: Randomized Metabolic Response Monitoring Trial in Patients With Suspected Recurrence of Glioblastoma FDOPA PET-CT
Brief Title: Response Monitoring Trial in Patients With Suspected Recurrence of Glioblastoma
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: PI left HMRI
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00009857; 121638 (Other: Principal Investigator); 1013-0158 (Other: HMRI IRB)
Record Dates: First submitted 2014-06-24; First posted 2014-06-27 (Estimated); Last update posted 2018-08-17 (Actual); Status verified 2018-08

CONDITIONS: Glioma; Glioblastoma; Glioblastoma Multiforme
Keywords: Glioma; Glioblastoma; Glioblastoma multiforme; GBM; Recurrence; PET; FDOPA
MeSH Terms: conditions — Glioma; Glioblastoma; Recurrence | interventions — fluorodopa F 18

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard diagnostics without PET (No Intervention): Standard of care brain imaging modalities, predominantly MRI
- FDOPA PET-CT (Experimental): PET-CT with administration of FDOPA as an experimental radiopharmaceutical. This arm includes standard of care imaging plus FDOPA PET-CT
  Interventions: Drug: FDOPA PET

INTERVENTIONS:
Drug: FDOPA PET — [18F]FDOPA radiopharmaceutical will be intravenousely injected for PET-CT scanning of the brain.
  Other Names: FDOPA PET-CT; Fluorine-18-L-dihydroxyphenylalanine; Fluorine-18-L-dihydroxyphenylalanine PET; Fluorine-18-L-dihydroxyphenylalanine PET-CT; [18F]FDOPA; [18F]FDOPA PET; [18F]FDOPA PET-CT
  Arms: FDOPA PET-CT

SUMMARY:
It was previously shown that [18F]Fluorodopa (FDOPA) PET imaging results in intended management changes in 41% of brain tumor patients. However, its impact on patient outcome defined as survival, costs, and/or quality of life has not been demonstrated. Regulatory agencies require randomized trials to determine the impact of PET on patient management and outcome. In this study we hypothesize that the addition of FDOPA PET will improve patient outcome by more accurately identifying presence or absence of tumor recurrence than conventional imaging.

DETAILED DESCRIPTION:
Malignant gliomas are aggressive primary brain tumors that almost always lead to rapid patient deterioration and death. Timely diagnosis of recurrent disease as well as accurate monitoring of therapeutic responses is critically important in glioblastoma patients.

Despite introduction of new treatment approaches patient prognosis is poor with less than half of the patients being progression-free during the first 6 months after diagnosis of disease recurrence (6-month-progression-free survival rates of 46%).

The current diagnostic standard of care for diagnosing and monitoring brain tumors is contrast-enhanced, multi-planar magnetic resonance imaging (MRI). However, the ability of MRI for early detection of disease recurrence or progression is limited. Moreover, determination of treatment responses is difficult since benign tissue changes after radiation and/or chemotherapy can have the appearance of tumor recurrence or progression on MRI. Positron emission tomography (PET) is an established imaging technique that utilizes small amounts of radioactivity attached to very minimal amounts of substances (tracers) that are injected via a hand or arm vein. These substances can track certain features of cancers that can be visualized by using the PET-CT scanner. For instance, a number of different PET-tracers have been used to study brain tumor metabolism and to detect primary or recurrent tumors. These include tracers of glucose ([18F]FDG) and amino acid metabolism (e.g., [11C] methionine and [18F]FDOPA). Metabolic imaging of brain tumors with amino acid analogues has advantages over FDG. Since FDG assess glucose metabolism and the normal brain consumes a lot of glucose it can be difficult to detect tumors against high glucose use of normal brain tissue. FDOPA has been successfully used clinically for many years. The advantage of FDOPA is that normal brain tissue consumes very little FDOPA. Thus, tumors can be seen easily against a low background activity.

FDOPA PET imaging detects brain tumors with a very high accuracy and affects the management of 40% of patients. However, its impact on patient outcome defined as survival, costs, and/or quality of life has not been demonstrated.

Randomized trials are needed to evaluate the impact of PET on patient management and outcome. We will determine this by randomizing patients with suspected recurrence of glioblastoma into those who are managed using conventional diagnostic imaging versus those who will receive conventional imaging plus FDOPA PET. Randomization is like flipping a coin. Patients will have a 50% chance to undergo standard imaging or standard imaging combined with FDOPA PET.

Approximately 25-40% of the patients with suspected tumor recurrence will have pseudo-progression on MRI (i.e., the images suggest that there is tumor recurrence when there is in fact no recurrence). These patients will have correctly negative FDOPA PET scans. In these patient initiation of treatment can be postponed. In contrast, patients with positive FDOPA PET scans will undergo some kind of treatment at the discretion of the treating physician (radiation therapy, chemotherapy or surgery). We will find out whether the management and treatment change that is based on FDOPA PET affects the survival of patients and affects the costs of caring for the patients.

ELIGIBILITY:
Inclusion Criteria:

* Suspected first recurrence of a glioblastoma tumor by clinical measures and/or MRI
* Age 18 and older

Exclusion Criteria:

* Breast feeding/ Pregnancy
* Severe psychiatric illness
* Primary diagnosis of a glioblastoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2014-05; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy compared to standard diagnostics without PET | 5 years
  Imaging findings will be validated by histopathology, clinical follow-up and/or repetitive imaging. If no histopathology within 3 months is available, clinical follow-up and imaging findings will be used for validation. If within 6 months of randomization no clinical progression nor progression on other imaging modalities is found, the patient will be rated as "no disease present at time of imaging".

SECONDARY OUTCOMES:
Impact of FDOPA PET on patient management | [ Time Frame: 7 years ]
  Overall and progression free survival will be assessed according to the standard of clinical care with a minimum follow-up time of two years after randomization. In this study protocol there are no pre-set follow-up algorithms, however in clinical routine a follow-up every three months is standard.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel Lee, MD, PhD, Principal Investigator — The Methodist Hospital Research Institute
Locations (1):
- Houston Methodist Research Institute PET Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No
No plan to share data.

REFERENCES:
- See also: Collaborator — https://clinicaltrials.gov/ct2/show/study?term=FDOPA&rank=10